Date: February 1st, 2022

## Study Protocol and Statistical Analysis Plan

| Study Title | A Novel, Non-pharmacological, Intervention for the |
|-----------------------|----------------------------------------------------|
| | Management of ADHD in Adolescents |
| Protocol ID | VIZO_004 |
| ClinicalTrials.gov ID | NCT05835336 |

| Device Name | VIZO Glasses |
|---|---|
| Objectives | To Assess the Efficacy and Safety of a Novel Device (VIZO Glasses) in the Management of ADHD in Adolescents. |
| Study Group Investigational Group | VIZO Glasses: Eyeglasses with personalized peripheral retinal stimuli |
| Key Eligibility Criteria | |
| Inclusion Criteria | <ul> <li>Documented history of primary ADHD diagnosis by certified clinicians</li> <li>Age 12-17 y</li> <li>Minimum total of 24 on the parent ADHD-IV Rating Scale (ADHD-RS)</li> <li>Written informed consent</li> <li>Able and willing to complete all required ratings and assessments</li> </ul> |
| Exclusion Criteria | <ul> <li>Any current psychiatric/neurological comorbidity (e.g., epilepsy, Autism, depression, TBI, etc.), other than ADHD</li> <li>ADHD Medications (stimulants, non-stimulants, other)</li> <li>Undergoing Neurofeedback, cognitive training</li> <li>Any other reason that, in the opinion of the investigator, prevents the participant from participating in the study</li> </ul> |
| Endpoints | |
| Primary | Primary Outcome Measure: Change in the ADHD Rating Scale (ADHD-RS) Parent-report Questionnaire - Total Score [Time Frame: Baseline, 2- month] The ADHD-RS is a parent report questionnaire that is used to aid in the diagnosis of ADHD in children ranging from ages 5- 17. The questionnaire contains 18 symptom items corresponding to the DSM-V criteria for ADHD. The parent rates each symptom item on a 4-point Likert scale ranging from 0 ('Never or Rarely') to 3 ('Very Often'). The total score goes from 0 up to 54. Higher scores mean more symptoms and higher ADHD impairments. |
| | Change in the ADHD Rating Scale (ADHD-RS) Parent-report Questionnaire - Inattention Subscale [Time Frame: Baseline, 2-month] The Inattention subscale of the ADHD-RS contains 9 symptom |

VIZO\_004 

items, that are designed to measure the child's attention level on tasks or play activities. The items are rated by the parent on a 4-point Likert scale ranging from 0 ('Never or Rarely') to 3 ('Very Often'). The total score goes from 0 up to 27. Higher scores mean more symptoms and higher ADHD impairments.

Change in the ADHD Rating Scale (ADHD-RS) Parent-report Questionnaire - Hyperactivity-Impulsivity Subscale [Time Frame: Baseline, 2-month]

The Hyperactivity-Impulsivity subscale of the ADHD-RS contains 9 symptom items, that are designed to measure the child's hyperactivity level and impulsivity level. The items are rated by the parent on a 4-point Likert scale ranging from 0 ('Never or Rarely') to 3 ('Very Often'). The total score goes from 0 up to 27. Higher scores mean more symptoms and higher ADHD impairments.

Change in Behavior Rating Inventory of Executive Function (BRIEF) - Metacognitive Index [Time Frame: Baseline, 2-month]

The Metacognition Index (MI) of the BRIEF reflects a child's ability to self-manage and monitor tasks cognitively. The subscale is composed of the Initiate, Working Memory, Plan/Organize, Organization of Materials, and Monitor scales of the BRIEF. It uses a Likert-type response format ranging from 1 to 3, where 1 is never, 2 is sometimes, and 3 is often. High scores indicate executive deficit.

## Secondary

Secondary Outcome Measures:

Clinical Global Impression-Improvement (CGI-I) [Time Frame: 2-month]

Based on an interview with the participant, the clinician rates the total improvement on a 7 point scale as follows: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.

Change in Behavior Rating Inventory of Executive Function (BRIEF) - Global Executive Composite [Time Frame: Baseline, 2-month]

The BRIEF is a standardized measure that captures views of

VIZO\_004 

| | executive functions or self-regulation in the everyday |
|---|---|
| | environment. The BRIEF is composed of 86 items, where each item is rated by the parent, using a 3-point Likert scale |
| | ranging from 1 ('Never') to 3 ('Often'). The Global Executive |
| | Composite (GEC) is an overarching summary score that |
| | incorporates all of the BRIEF clinical scales. High scores |
| | indicate executive deficit. |
| Other Outcomes | Adverse events will be monitored and documented. |
| Follow-up Visits Schedule | This was a two-month, open-label study in which eligible ADHD-diagnosed adolescents were provided with a pair of VIZO- |
| | Glasses featuring a personalized visual stimuli pattern for each |
| | participant. A baseline assessment of the participants' ADHD |
| | clinical profile pre-intervention included the ADHD-RS and the |
| | Behavior Rating Inventory of Executive Function (BRIEF) |
| | questionnaires. In addition, participants completed the |
| | Conners' Continuous Performance Test-3 (CPT-3). Optical |
| | centration parameters and demographic information were |
| | collected for each participant. Participants were then invited to |
| | complete a personalization process in which they were fitted |
| | with personalized VIZO-glasses. Participants were instructed to |
| | wear their Vizo-glasses for at least two hours daily for two |
| | months. A follow-up assessment at the end of the intervention |
| | re-assessed ADHD performance on the ADHD-RS and BRIEF |
| | questionaries. In addition, participants completed the CPT-3 |
| | test while wearing their VIZO-glasses. The Clinical Global |
| | Impression-Improvement (CGI-I) rating scale was administered |
| | by a clinician. |
| Sample Size | Given the exploratory nature of the study, the sample size was |
| | chosen to be sufficiently large to detect significant within |
| | subject effects of at least 0.5 (Cohen's D) for a 2-Tailed test, at |
| | anlpha-0.05 with a power of 80%. |
| Analysis Plan | Paired samples t-tests will be used to test the effect of the |
| • | VIZO-glasses intervention, comparing the baseline and end-of- |
| | intervention performances. No corrections for multiple testing |
| | will be applied due to the exploratory nature of the study. The |
| | safety analysis will include all available data on the intent-to- |
| | treat (ITT) population. |
| | 1 |

VIZO\_004 